CLINICAL TRIAL: NCT06026189
Title: Safely Reduce Cystoscopic Evaluations for Hematuria Patients
Acronym: SeARCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, J.L. Boormans, MD PhD, Professor, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Erasmus MC
Record Dates: First submitted 2023-08-01; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Hematuria; Urothelial Neoplasm; Urothelial Carcinoma; Bladder Cancer
Keywords: Urinary biomarker; Hematuria; Urothelial Carcinoma; Bladder Cancer
MeSH Terms: conditions — Hematuria; Carcinoma, Transitional Cell; Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: A multicenter, stepped wedge cluster randomized trial
Masking Description: This is a stepped wedge cluster randomized clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care-as-usual (No Intervention): In the ''care-as-usual'' arm, all patients undergo 'care-as-usual', i.e. a cystoscopy and upper tract imaging (ultrasound or CT-scan)
- 'Urine-first' strategy (Experimental): In the intervention arm, the urine test is used to triage patients for a diagnostic workup ('urine-first' strategy). Only patients with an abnormal test result undergo cystoscopy and upper tract imaging.
  Interventions: Diagnostic Test: urine-first strategy

INTERVENTIONS:
Diagnostic Test: urine-first strategy — Only patients with an abnormal urine test result undergo a diagnostic workup, i.e. cystoscopy and upper-tract imaging.
  Arms: 'Urine-first' strategy

SUMMARY:
The SeARCH-trial assess the clinical impact of a molecular urine test as a 'urine-first' strategy in the diagnostic workup of patients presenting with microscopic hematuria.

DETAILED DESCRIPTION:
Microscopic hematuria (MH) can be a sign of an underlying disease, including malignancy of the urinary tract, and is reason for referral to a urology clinic. The current standard diagnostic workup for MH patients includes visual inspection of the bladder by cystoscopy and upper tract imaging to rule out the presence of a tumor in the urinary tract. However, the a priori risk of cancer in patients with MH is only 2-5%. Consequently, 95% of MH patients unnecessarily undergo invasive procedures, which are: I) uncomfortable and stressful for patients, II) has a significant impact on limited available (financial) resources and III) a CT scan is accompanied by exposure to ionizing radiation.

Previously we developed a molecular urine assay to detect urinary tract cancer in hematuria patients that had robust diagnostic performance; a negative predictive value >99%, sensitivity, and specificity >90%. The SeARCH-trial evaluates the clinical impact of a urine assay as a 'urine-first' strategy, meaning that only patients with an abnormal urine test results undergo invasive diagnostics. In this multicenter stepped-wedge cluster randomized trial we compare clinical outcomes by using a 'urine-first' strategy to 'care-as-usual', which is a cystoscopy and upper tract imaging in all patients presenting with MH. In addition, we assess patients' preferences, patients reported outcome measurements, and healthcare costs to show that a 'urine-first' strategy improves patients' quality of life and results in a more appropriate use of limited available resources.

ELIGIBILITY:
Inclusion Criteria:

* Microscopically confirmed microscopic hematuria of voided urine defined as ≥3 erythrocytes per high power field
* Male patients ≥40 years
* Female patients ≥50 years

Exclusion Criteria:

* History of urothelial bladder- or urinary tract cancer
* Presence of macroscopic (visible) hematuria
* Woman who is or may be pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
The primary aim of the SeARCH-trial is to assess the clinical impact of implementing a molecular urinary assay as a 'urine-first' strategy, in the diagnostic workup of patients presenting with microscopic hematuria. | 1 year
  The net benefit is defined as the proportion of patients who were diagnose with urinary tract cancer within 1 year after initial diagnostic work-up in the population (true positives) subtracted by the proportion of patients that underwent diagnostic evaluations without an abnormal finding (false positives). The latter is multiplied by the decision threshold, which represents the estimated harms of the diagnostic intervention, such as patients' burden and use of available resources, against the harms of an outcome event, i.e. missing a urinary tract tumor.

SECONDARY OUTCOMES:
The number of cystoscopies and upper tract imaging modalities (CT or ultrasound) when using a 'urine-first' strategy versus 'care-as-usual' | 1 year
Cost-effectiveness analysis | Questionnaires are administered at baseline, 3, 6, and 12 months.
  This will be performed according to the Dutch guideline by administering validated questionnaires.
Patient reported outcome measurements (PROMs) | Questionnaires are administered at baseline, 3, 6, and 12 months.
  Patient-reported outcome measurements (PROMs) are assessed for patients undergoing cystoscopy and urine collection.

CONTACTS AND LOCATIONS:
Locations (1):
- SeARCH-trial Pijpers, Rotterdam, Netherlands